CLINICAL TRIAL: NCT01206491
Title: Development of Intervention Model for Osteoporosis and Fall Prevention in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Ling Tsai, Social Work Office
Other Study IDs: 99035
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Department of Chronic Disease and Health Promotion of World Health Organization listed eight classes of chronic disease which will be important globally in the future. And the sixth class is "Chronic Rheumatic Condition", which includes rheumatic arthritis, osteoarthritis, osteoporosis, spinal disorders and severe limb trauma. Obviously the osteoporosis is a globally important health topic.

Osteoporosis draws more and more attention, because osteoporosis has various influences, for example, (1) psychologically impact which occurs frequently in many chronic diseases, such as depression will appear evidently in patients with osteoporosis (2) patients with osteoporosis often lose their social role (3) osteoporosis might induce pain and limitation of body function (4) osteoporosis increases greatly the possibility of fracture. Osteoporosis will induce adverse outcomes, such as the fall of life quality, the increase of morbidity and mortality, as well as the increased abuse of medical service. In this project, the investigators will set up the intervention model for prevention of osteoporosis as well as falls.

In this project, the investigators will recruit patients form outpatient services at WanFang Hospital. Through the collection of baseline data from questionnaire and bone density measurement, the investigators can clarify the risk of osteoporosis and falls in studied patients. By using double-blind randomized design, the patients will be collected to either one of intervention and control group. After eight weeks of intervention programs, the investigators will follow on both groups to understand the effect of this program and to increase the bone density of intervention group. The hospital or the Health center might take the outcome to be the reference of taking care the Osteoporosis.

DETAILED DESCRIPTION:
Department of Chronic Disease and Health Promotion of World Health Organization listed eight classes of chronic disease which will be important globally in the future. And the sixth class is "Chronic Rheumatic Condition", which includes rheumatic arthritis, osteoarthritis, osteoporosis, spinal disorders and severe limb trauma. Obviously the osteoporosis is a globally important health topic.

Osteoporosis draws more and more attention, because osteoporosis has various influences, for example, (1) psychologically impact which occurs frequently in many chronic diseases, such as depression will appear evidently in patients with osteoporosis (2) patients with osteoporosis often lose their social role (3) osteoporosis might induce pain and limitation of body function (4) osteoporosis increases greatly the possibility of fracture. Osteoporosis will induce adverse outcomes, such as the fall of life quality, the increase of morbidity and mortality, as well as the increased abuse of medical service. In this project, we will set up the intervention model for prevention of osteoporosis as well as falls.

In this project, we will recruit patients form outpatient services at WanFang Hospital. Through the collection of baseline data from questionnaire and bone density measurement, we can clarify the risk of osteoporosis and falls in studied patients. By using double-blind randomized design, the patients will be collected to either one of intervention and control group. After eight weeks of intervention programs, we will follow on both groups to understand the effect of this program and to increase the bone density of intervention group. The hospital or the Health center might take the outcome to be the reference of taking care the Osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* the risk of osteoporosis
* the risk of falls

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we will recruit patients form outpatient services at WanFang Hospital or the people who live near WanFang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2010-09; Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ling Tsai, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan